CLINICAL TRIAL: NCT03297333
Title: Effects of Exercise Mode on Cardiac Fat and Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid/19
Sponsor: Southern Illinois University Edwardsville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1208-4C-1
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: Obesity; Exercise; Cardiac Fat; Cardiac Magnetic Resonance; Vascular Health
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance training group (Experimental): Resistance training will consist of a supervised circuit training 3 sessions/week for approximately 45-50 min/session. The circuit will include 7 strength exercises engaging the major muscle groups (leg press, rows, back squats, weighted crunches, deadlifts, bench press, and squat jumps with weights). The participants will perform 3 sets of 10 repetitions with resting periods of 30 seconds between exercises, and 2 minutes between sets. The overall OMNI-Resistance Exercise Scale per set will range between 8-10. Heart rate and exercise energy expenditure during the workout will be monitored. The load will be changed depending on the participants' perception when needed. In addition, the intensity will be monitored assessing Lactate concentrations at baseline and at the end of each session. Circuit will be repeated until meeting the targeted exercise energy expenditure of 450-500 kcal/session.
  Interventions: Other: Resistance training
- Aerobic interval training group (Experimental): Aerobic interval will consist of a supervised aerobic interval training sessions 3 times/week. Duration will range between 45-50 min/session depending on the exercise energy expenditure. Each interval will have a total duration of 5 min, and it will be divided into 2 periods. The first period will consist of 3 minutes of high-intensity activity, and the second period the intensity will be reduced for 2 minutes. The speed/incline will be changed depending on the participants' heart rate and perception using the Borg's rating of perceived exertion as needed. Heart rate and exercise energy expenditure during the workout will be monitored. Intensity will be monitored assessing Lactate concentrations at the end of each session. Intervals will be repeated until meeting the targeted exercise energy expenditure (450-500 kcal/session).
  Interventions: Other: Aerobic interval training
- Control group (No Intervention): Participants in the control group will not participate in the training programs.

INTERVENTIONS:
Other: Resistance training — The resistance training group
  Arms: Resistance training group
Other: Aerobic interval training — The aerobic interval training group
  Arms: Aerobic interval training group

SUMMARY:
The overall goal of this project is to study the effects of exercise energy expenditure matched vigorous dynamic resistance training and aerobic training on cardiac fat, and its relationship to cardiac function and geometry using cardiac Magnetic Resonance Imaging.

DETAILED DESCRIPTION:
Exercise-induced weight-loss is one of the most common strategies for reducing excess fat in overweight and obese individuals. Although vigorous intensity may be more favorable promoting positive cardiac adaptations compared to low-moderate intensity, evidence of the positive effects of different exercise modes needs to be explored to allow for realistic comparisons with other strategies. Research using cardiac Magnetic Resonance Imaging that compares the effects of different modes of exercise - matched by exercise energy expenditure - on epicardial adipose tissue and paracardial adipose tissue, and how these interventions modify cardiac function and geometry have not been previously explored in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* Caucasian
* BMI >30 kg/m2 and < 39.9 kg/m2

Exclusion Criteria:

* Known cardiovascular, metabolic, pulmonary disease or conditions
* Muscular-skeletal injuries
* Taking medications that affect endocrine or cardiovascular function
* Hypertension
* Being engaged in low intensity strength training more than two times per week or moderate-high intensity of any type of frequency
* Being pregnant
* Cigarette smoking
* Having non-removable pieces or devices incompatible with DXA and CMR assessment.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Changes in Epicardial adipose tissue (EAT) | 2 assessment points: at baseline and week 4
  EAT will be measured using cardiac Magnetic Resonance
Changes in Vascular Health | 2 assessment points: at baseline and week 4
  Atrial stiffness will be measured using a pulse wave analysis

SECONDARY OUTCOMES:
Changes in Paracardial adipose tissue (PAT) | 2 assessment points: at baseline and week 4
  PAT will be measured using cardiac Magnetic Resonance
Changes in Body Composition | 2 assessment points: at baseline and week 4
  Body composition will be measured using dual-energy x-ray absorptiometry
Changes in Cardiorespiratory Function | 2 assessment points: at baseline and week 4
  Cardiorespiratory Function will be measured on a treadmill with a metabolic cart
Changes in Muscular Strength | 2 assessment points: at baseline and week 4
  Muscular Strength will be assessed by 1 repetition maximum (1RM) test

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Southern Illinois University of Edwardsville
Locations (1):
- Southern Illinois University of Edwardsville, Edwardsville, Illinois, United States